CLINICAL TRIAL: NCT04503265
Title: A Phase I/II, Open Label, Multi-center, Non-randomized Dose Escalation and Dose Expansion Study of AMXI-5001 in Patients With Advanced Malignancies
Brief Title: A Trial of AMXI-5001 for Treatment in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AtlasMedx, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS-101
Record Dates: First submitted 2020-07-23; First posted 2020-08-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Neoplasm; Breast Cancer; Ovarian Cancer; Homologous Recombination Deficiency; Prostate Cancer; Pancreatic Cancer
Keywords: Breast; Ovarian; Prostate; Pancreatic; Refractory; Cancer; Malignancy; BRCA; HRD; AMXI-5001; Progression; PARP Inhibitor; Microtubule inhibitor
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Neoplasms; Disease Progression | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AMXI-5001 Treatment (Experimental): Single Arm Study, all participants will receive AMXI-5001.
  Interventions: Drug: AMXI-5001:Dose Escalation Phase I; Drug: AMXI-5001:Dose Expansion Phase II

INTERVENTIONS:
Drug: AMXI-5001:Dose Escalation Phase I — Phase I will enroll up to 70 participants to identify the Recommended Phase II daily dose in the treatment of various cancers and to characterize the safety, pharmacology, and clinical efficacy of AMXI-5001. AMXI-5001 is administered orally twice daily, with food. AMXI-5001 is administered weekly on a continuous 7-day schedule. Each cycle is 28 days.
  Other Names: Phase I; Dose Escalation
Drug: AMXI-5001:Dose Expansion Phase II — Phase II will enroll up to 52 study participants to further characterize the safety, pharmacology, and clinical efficacy of AMXI-5001. AMXI-5001 is administered orally twice daily, with food. AMXI-5001 is administered weekly on a continuous 7-day schedule. Each cycle is 28 days.
  Other Names: Phase II; Dose Expansion

SUMMARY:
ATLAS-101 is a Phase I/II clinical trial of AMXI-5001 in adult participants with advanced malignancies who have previously failed other therapies. The study has two phases. The purpose of Phase I (Dose Escalation) is to confirm the appropriate treatment dose and Phase II (Dose Expansion) is to characterize the safety and efficacy of AMXI-5001.

DETAILED DESCRIPTION:
AMXI-5001 is an orally available dual PARP (poly adenosine diphosphate [ADP] ribose polymerase) and microtubule polymerization inhibitor. ATLAS-101 is a Phase I/II, open label, multi-center, non-randomized Dose Escalation and Dose Expansion study in participants with advanced malignancies. Study enrollment is approximately 122 participants. All participants receive oral AMXI-5001, twice daily, as monotherapy. Following Phase I (Dose Escalation) to identify the Maximum Tolerated Dose and the Recommended Dose for use in Phase II, additional participants will be enrolled into the Dose Expansion Phase to further characterize the safety, pharmacology, and clinical efficacy of AMXI-5001.

ELIGIBILITY:
Inclusion Criteria (Key Factors):

1. Has pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following:

   1. Patient is intolerant of existing therapy(ies) known to provide clinical benefit for their condition
   2. Malignancy is refractory to existing therapy(ies) known to potentially provide clinical benefit
   3. Malignancy has progressed after standard therapy
2. Has evaluable or measurable tumor(s) in dose escalation by standard radiological and/or laboratory assessments as applicable to their malignancy.
3. Eastern Co-operative Oncology Group (ECOG) PS 0-1
4. Participant must be 18 years of age or older
5. Able to understand and sign consent

Exclusion Criteria (Key Factors):

1. Receiving cancer treatment at the time of enrollment
2. Any clinically significant disease or condition affecting a major organ system
3. Significant cardiovascular disease or electrocardiogram (ECG) abnormalities
4. Use of a strong inhibitor or inducer of CYP3A4 within 7 days prior to start of study therapy and throughout the study (e.g., some antibiotics, antifungals, anticonvulsants, grapefruit)
5. Has had a previous (within 2 years) or has a current malignancy other than the target cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) | Approximately 12 months
  The highest dose is defined at which no more than 1 of 6 evaluable participants has had a Dose Limiting Toxicity (DLT) according to NCI CTCAE V5.0 criteria and determination by Investigator and Data and Safety Monitoring Committee.
Determine the Recommended Phase 2 Dose (RP2D) for AMXI-5001 as monotherapy | Approximately 12 months
  The RP2D is based upon the review of all available data including safety, pharmacokinetic, preliminary anti-tumor activity, and MTD.
Characterize safety profile of AMXI-5001 | Approximately 24 months
  The safety profile of AMXI-5001 is defined by the incidence of treatment emergent adverse events, laboratory abnormalities, and ECG measurements.

SECONDARY OUTCOMES:
Measure concentration of AMXI-5001 in plasma samples | Approximately 24 months
  Concentrations of AMXI-5001 in plasma samples at different time points are measured. Standard pharmacokinetic parameters are calculated.
Determine change in anti-tumor activity following administration of AMXI-5001 | Approximately 24 months
  Overall Survival (OS), Objective Response Rate (ORR), Duration of Response (DOR), and Progression-free Survival (PFS) are assessed by RECIST V1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Study Director — AtlasMedx, Incorporated
Locations (4):
- United States (4):
  - University of California, Los Angles (UCLA) Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Johns Hopkins, Baltimore, Maryland
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemjabbar-Alaoui H, Peto CJ, Yang YW, Jablons DM. AMXI-5001, a novel dual parp1/2 and microtubule polymerization inhibitor for the treatment of human cancers. Am J Cancer Res. 2020 Aug 1;10(8):2649-2676. eCollection 2020. PMID 32905466
- See also: Citation — https://pubmed.ncbi.nlm.nih.gov/32905466/